CLINICAL TRIAL: NCT03973749
Title: Effects of a High or Low Salycilate Diet on Urinary Leucotriene E4 Levels and Clinical Features in Patients With Aspirin Exacerbated Respiratory Disease
Brief Title: Effects of a High or Low Salycilate Diet on Urinary LTE4 and Clinical Features in AERD
Acronym: AERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Marcos Alejandro Jimenez Chobillon, Professor, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: C13-17
Record Dates: First submitted 2019-02-06; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Aspirin-exacerbated Respiratory Disease; Aspirin-Sensitive Asthma With Nasal Polyps; Samter's Syndrome; Widal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Low salycilate diet on day one and High salycilate diet on day 7
  Interventions: Other: Low salycilate diet
- Group 2 (Experimental): High salycilate diet on day one and Low salycilate diet on day 7
  Interventions: Other: Low salycilate diet

INTERVENTIONS:
Other: Low salycilate diet — Each arm of the experimental group will be exposed to low and high concentrations of dietary salycilates and urinary LTE4, FEV1, FVC, FEV1/FVC and total inspiratory nasal resistance will be measured at basal level and then two hours after each of the 3 daily meals.
  Other Names: High salycilate diet

SUMMARY:
On day one, two groups of nine patients each will respectively recieve the tree daily meals (breakfast, Lunch and dinner) in a controled clinical setting. Group 1 will recieve a low-salycilate diet, and group 2 a high-salycilate diet. Two hours after each meal, urinary Leucotriene E4, FEV1, FVC, FEV1/FVC and total nasal resistance will be measured. On day 7, after clearance time, group 1 will recieve high-salycilate diet and group 2 low salycilate diet and the same measurements will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Aspirin exacerbated respiratory disease.
* Controled asthma
* No actual systemic corticosteroid treatment
* No antileucotriene treatment.

Exclusion Criteria:

* Patients who do not complete both phases of the study
* Patients unable to perform adecuate spyrometric testing
* Patients who present severe asthmatic reactions with high salycilate foods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Urinary concentration of Leucotriene E4 (LTE4) | Baseline-4-8-12 hours in day one and Baseline-4-8-12 hours in day 7
  pg/ml of creatinine

SECONDARY OUTCOMES:
Change from baseline in Expiratory Volume in 1 second (FEV-1) | Baseline-4-8-12 hours and Baseline-4-8-12 hours in day 7
  Percentage of referenced value
Change from baseline in Vital Capacity (FVC) | Baseline-4-8-12 hours and Baseline-4-8-12 hours in day 7
  Percentage of referenced value
Change from baseline in the Relationship between FEV1/FVC | Baseline-4-8-12 hours and Baseline-4-8-12 hours in day 7
  Percentage of referenced value
Change from baseline in the total nasal resistance obtained by rhinometry | Baseline-4-8-12 hours and Baseline-4-8-12 hours in day 7
  pascals/cm3/sec

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No